CLINICAL TRIAL: NCT01815918
Title: The Effect of Low Dose Corticosteroids on Perioperative Markers of Thrombosis and Fibrinolysis in Total Knee Arthroplasty
Brief Title: Effect of Low Dose Corticosteroids on Perioperative Markers of Thrombosis and Fibrinolysis in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-054
Record Dates: First submitted 2013-02-12; First posted 2013-03-21 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Total Knee Arthroplasty
Keywords: Orthopedic Procedures; Prostheses and Implants; Joint Prosthesis; Knee Prosthesis; Arthroplasty, Knee; Thromboembolism; Inflammation; B-Cell Differentiation Factor-2; Differentiation Factor-2, B-Cell; B-Cell Stimulatory Factor-2; BSF-2; IFN-beta 2; MGI-2; Interleukin-6 (IL-6); Steroids; Pregnenediones; Hydrocortisone; Physiological Effects of Drugs; Therapeutic Uses
MeSH Terms: conditions — Thromboembolism; Inflammation | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients receive a saline placebo before surgery, 8 hours after the first dose and 16 hours after the first dose.
  Interventions: Drug: Placebo
- Treatment (Active Comparator): Patients receive 3 100 mg of hydrocortisone: prior to surgery, 8 hours after the first dose and 16 hours after the first dose.
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Patients randomized to treatment arm will three doses of 100 mg of hydrocortisone at the following times: prior to surgery, 8 hours after the first dose and 16 hours after the first dose.
  Other Names: Ala-Cort; Ala-Scalp HP; Anusol HC; Aquanil HC; Beta HC; Cetacort; Colocort; Corta-Cap
  Arms: Treatment
Drug: Placebo — Patients receive placebo prior to surgery, 8 hours after the first dose and 16 hours after the first dose.
  Arms: Placebo

SUMMARY:
One postoperative complication following unilateral or bilateral total knee arthroplasty is thrombosis (blood clot formation). In this prospective, double-blinded randomized controlled clinical trial, researchers are investigating the effect of steroids on biochemical markers of thrombosis. Furthermore, elevated cellular markers of thrombosis (specifically IL-6) have been linked to postoperative depression following total knee arthroplasty surgery. Hence the investigators are also checking if use of hydrocortisone, a steroid, may help reduce the incidence of postoperative depression.

Other studies have shown that surgery causes some reaction in the body that is consistent with inflammation. When the inflammation is extensive, it may affect different parts of the body. It may also lead to clotting disorders and result in blood clots. In a previous study by this principal investigator (see reference 22, "Use of low-dose steroids in decreasing cytokine release during bilateral total knee arthroplasty"), hydrocortisone was administered over 24 hours following surgery to patients who underwent bilateral total knee arthroplasty. The investigator found lower levels of cellular markers consistent with inflammation (specifically the protein, IL-6). Steroid use also showed additional benefits, such as decreased pain and better range of motion at the knee.

In this study, investigators recruit patients undergoing total knee arthroplasty surgery. Patients are randomized to receive three 100 mg doses of hydrocortisone or three doses of a saline placebo. In addition to analyzing patients' blood samples for hydrocortisone's effect on clotting factors (i.e. IL-6), investigators record patients' pain scores and patients' oral analgesic use. To assess patients' well-being, patients are contacted one month and 3 months following their surgeries and administered the Patient Health Questionnaire (see reference 23, "The PHQ-9: validity of a brief depression severity measure.") arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing unilateral or bilateral total knee replacement
* Age 50-90

Exclusion Criteria:

* All patients on steroid therapy regardless of dose or duration of treatment or those requiring stress-dose steroids preoperatively
* Patients who are smokers
* Patients under 50 years of age
* Patients over 90 years of age
* Patients with diabetes
* Patients with a prior history of corticosteroid intolerance
* Patients with previous complications of steroid use

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kethy Jules-Elysée, M.D., Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Boermeester MA, van Leeuwen PA, Coyle SM, Wolbink GJ, Hack CE, Lowry SF. Interleukin-1 blockade attenuates mediator release and dysregulation of the hemostatic mechanism during human sepsis. Arch Surg. 1995 Jul;130(7):739-48. doi: 10.1001/archsurg.1995.01430070061012. PMID 7611862
- [Background] Busso N, Belin D, Failly-Crepin C, Vassalli JD. Plasminogen activators and their inhibitors in a human mammary cell line (HBL-100). Modulation by glucocorticoids. J Biol Chem. 1986 Jul 15;261(20):9309-15. PMID 3087993
- [Background] Collen D, Hoylaerts MF. Relationship between inflammation and venous thromboembolism as studied by microparticle assessment in plasma. J Am Coll Cardiol. 2005 May 3;45(9):1472-3. doi: 10.1016/j.jacc.2005.02.029. No abstract available. PMID 15862421
- [Background] Cremeans-Smith JK, Soehlen S, Greene K, Alexander T, Delahanty DL. In-hospital levels of C-reactive protein and IL-6 predict post-operative depressive symptoms among patients undergoing total knee replacement surgery. Brain Behav Immun. 2009 Nov;23(8):1096-103. doi: 10.1016/j.bbi.2009.06.148. Epub 2009 Jun 24. PMID 19559081
- [Background] Fox EA, Kahn SR. The relationship between inflammation and venous thrombosis. A systematic review of clinical studies. Thromb Haemost. 2005 Aug;94(2):362-5. doi: 10.1160/TH05-04-0266. PMID 16113826
- [Background] Hogevold HE, Hoiseth A, Reikeras O. Effect of high-dose corticosteroids on the incidence of deep vein thrombosis after total hip replacement. Arch Orthop Trauma Surg. 1991;111(1):29-31. doi: 10.1007/BF00390189. PMID 1722989
- [Background] Jansen NJ, van Oeveren W, van den Broek L, Oudemans-van Straaten HM, Stoutenbeek CP, Joen MC, Roozendaal KJ, Eysman L, Wildevuur CR. Inhibition by dexamethasone of the reperfusion phenomena in cardiopulmonary bypass. J Thorac Cardiovasc Surg. 1991 Oct;102(4):515-25. PMID 1656149
- [Background] Levi M, Cromheecke ME, de Jonge E, Prins MH, de Mol BJ, Briet E, Buller HR. Pharmacological strategies to decrease excessive blood loss in cardiac surgery: a meta-analysis of clinically relevant endpoints. Lancet. 1999 Dec 4;354(9194):1940-7. doi: 10.1016/S0140-6736(99)01264-7. PMID 10622296
- [Background] Levi M, van der Poll T. Two-way interactions between inflammation and coagulation. Trends Cardiovasc Med. 2005 Oct;15(7):254-9. doi: 10.1016/j.tcm.2005.07.004. PMID 16226680
- [Background] Medcalf RL, Van den Berg E, Schleuning WD. Glucocorticoid-modulated gene expression of tissue- and urinary-type plasminogen activator and plasminogen activator inhibitor 1 and 2. J Cell Biol. 1988 Mar;106(3):971-8. doi: 10.1083/jcb.106.3.971. PMID 3126194
- [Background] Medcalf RL, Kruithof EK, Schleuning WD. Plasminogen activator inhibitor 1 and 2 are tumor necrosis factor/cachectin-responsive genes. J Exp Med. 1988 Aug 1;168(2):751-9. doi: 10.1084/jem.168.2.751. PMID 3137305
- [Background] Nilsson T, Carlsson J, Sundqvist G. Inactivation of key factors of the plasma proteinase cascade systems by Bacteroides gingivalis. Infect Immun. 1985 Nov;50(2):467-71. doi: 10.1128/iai.50.2.467-471.1985. PMID 3902645
- [Background] Parvizi J, Mui A, Purtill JJ, Sharkey PF, Hozack WJ, Rothman RH. Total joint arthroplasty: When do fatal or near-fatal complications occur? J Bone Joint Surg Am. 2007 Jan;89(1):27-32. doi: 10.2106/JBJS.E.01443. PMID 17200306
- [Background] Pulido L, Ghanem E, Joshi A, Purtill JJ, Parvizi J. Periprosthetic joint infection: the incidence, timing, and predisposing factors. Clin Orthop Relat Res. 2008 Jul;466(7):1710-5. doi: 10.1007/s11999-008-0209-4. Epub 2008 Apr 18. PMID 18421542
- [Background] Reikeras O, Clementsen T. Thrombosis markers in hip versus knee arthroplasty: a pilot study. J Orthop Surg (Hong Kong). 2009 Dec;17(3):291-5. doi: 10.1177/230949900901700309. PMID 20065366
- [Background] Sharrock NE, Go G, Sculco TP, Salvati EA, Westrich GH, Harpel PC. Dose response of intravenous heparin on markers of thrombosis during primary total hip replacement. Anesthesiology. 1999 Apr;90(4):981-7. doi: 10.1097/00000542-199904000-00009. PMID 10201667
- [Background] van der Poll T, Levi M, Hack CE, ten Cate H, van Deventer SJ, Eerenberg AJ, de Groot ER, Jansen J, Gallati H, Buller HR, et al. Elimination of interleukin 6 attenuates coagulation activation in experimental endotoxemia in chimpanzees. J Exp Med. 1994 Apr 1;179(4):1253-9. doi: 10.1084/jem.179.4.1253. PMID 8145042
- [Background] van Deventer SJ, Buller HR, ten Cate JW, Aarden LA, Hack CE, Sturk A. Experimental endotoxemia in humans: analysis of cytokine release and coagulation, fibrinolytic, and complement pathways. Blood. 1990 Dec 15;76(12):2520-6. PMID 2124934
- [Background] van Giezen JJ, Chung-A-Hing JE, Vegter CB, Bouma BN, Jansen JW. Fibrinolytic activity in blood is distributed over a cellular and the plasma fraction which can be modulated separately. Thromb Haemost. 1994 Dec;72(6):887-92. PMID 7740459
- [Background] Voshaar RC, Banerjee S, Horan M, Baldwin R, Pendleton N, Proctor R, Tarrier N, Woodward Y, Burns A. Predictors of incident depression after hip fracture surgery. Am J Geriatr Psychiatry. 2007 Sep;15(9):807-14. doi: 10.1097/JGP.0b013e318098610c. Epub 2007 Aug 13. PMID 17698601
- [Background] Wagner DD, Burger PC. Platelets in inflammation and thrombosis. Arterioscler Thromb Vasc Biol. 2003 Dec;23(12):2131-7. doi: 10.1161/01.ATV.0000095974.95122.EC. Epub 2003 Sep 18. PMID 14500287
- [Background] Jules-Elysee KM, Lipnitsky JY, Patel N, Anastasian G, Wilfred SE, Urban MK, Sculco TP. Use of low-dose steroids in decreasing cytokine release during bilateral total knee replacement. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):36-40. doi: 10.1097/AAP.0b013e31820306c5. PMID 21455087
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Derived] McLawhorn AS, Poultsides LA, Sakellariou VI, Kunze KN, Fields KG, Jules-Elysee K, Sculco TP. Low-Dose Perioperative Corticosteroids Can Be Administered Without Additional Morbidity in Patients Undergoing Bilateral Total Knee Replacement: A Retrospective Follow-up Study of a Randomized Controlled Trial. HSS J. 2022 Feb;18(1):48-56. doi: 10.1177/15563316211006098. Epub 2021 Apr 9. PMID 35087332
- See also: This is a link to the Hospital for Special Surgery home page. — http://www.hss.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Treatment
Started | 30 | 30
Completed | 12 | 11
Not Completed | 18 | 19
Not completed — Patient samples not analyzable | 3 | 4
Not completed — Lack of Efficacy | 15 | 15

BASELINE CHARACTERISTICS:
Population: Unilateral Total Knee Replacement
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Treatment | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8) | 68 (6) | 67 (7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 8 | 8 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Prothrombin Fragment (PF1.2), a Marker of Thrombin Generation
Description: Study patients received 100 mg of intravenous hydrocortisone 2 h prior to surgery, and controls received normal saline. Blood samples, drawn pre-incision and at 4 h post tourniquet release, were assayed for PF1.2 and PAP
Time Frame: Baseline and up to 4 hours following surgery
Measure: Mean (Standard Deviation); unit: pMol/L
Arm/Group | Placebo | Treatment
Number analyzed (Participants) | 12 | 11
pMol/L
  Baseline | 263.6 (158.6) | 266.5 (146.9)
  4s | 935.8 (331.9) | 615.9 (357.7)

2. Primary Outcome: Plasmin-alpha-2-antiplasmin Complex (PAP), a Marker of Fibrinolysis
Description: as for outcome 1
Time Frame: Baseline and up to 4 hours following surgery
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Placebo | Treatment
Number analyzed (Participants) | 12 | 11
ug/L
  Baseline | 623.3 (324.8) | 808.4 (372.1)
  4 hs | 1086.8 (536.3) | 1638.6 (823.2)

3. Secondary Outcome: Hydrocortisone's Effect on Depression
Description: Elevated IL-6 has been linked to post-operative depression following total knee replacement surgery. Patients will be administered the patient health questionnaire (PHQ-9) one month and 3 months following surgery to assess their well-being.
Time Frame: one month and up to 3 months following surgery
Population: Outcome could not be analyzed because patients could not be reached to collect data at one month and up to 3 months following surgery.
Groups:
- Placebo; Treatment: Data was not collected
Arm/Group | Placebo | Treatment
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pain Scores and Opioid Consumption
Description: Pain scores (rated on a scale of 0-10) will be taken throughout study participation. We will also record analgesic use to see if patients who received hydrocortisone needed fewer pain killers to control their postoperative pain.
Time Frame: one month and up to 3 months following surgery
Population: as for outcome 3
Arm/Group | Placebo | Treatment
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Blinding Assessment
Description: Throughout each patient's study participation, the patient and the data collector will be asked to guess their treatment status. This helps ascertain if there is an association between blinding status, treatment effect and the depression measure.
Time Frame: one month and up to 3 months following surgery
Population: as for outcome 3
Arm/Group | Placebo | Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Treatment
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes